CLINICAL TRIAL: NCT03501628
Title: The Effects of Different Protein and Amino Acid Supplements of Muscle Hypertrophy After 12 Weeks of Resistance Exercise in Untrained Men
Brief Title: Leucine or Protein Supplementation and Resistance Training
Acronym: MPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Michael Roberts, Associate Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-320 MR 1508
Record Dates: First submitted 2017-08-31; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Skeletal Muscle
MeSH Terms: interventions — Leucine; maltodextrin; Whey

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): 2 servings daily
  Serving information:
  * 204 kcal
  * 2.8 g fat
  * 44.4 g carbohydrate
  * 0.4 g protein (0 g L-leucine)
  Interventions: Dietary Supplement: Placebo
- L-leucine + maltodextrin (Experimental): 2 servings daily
  Serving information:
  * 200 kcal
  * 2.0 g fat
  * 43.1 g carbohydrate
  * 2.8 g protein (2.8 g L-leucine)
  Interventions: Dietary Supplement: L-leucine + maltodextrin
- Whey protein concentrate (Experimental): 2 servings daily
  Serving information:
  * 184 kcal
  * 3.5 g fat
  * 12 g carbohydrate
  * 26.3 g protein (2.8 g L-leucine)
  Interventions: Dietary Supplement: Whey protein concentrate
- Hydrolyzed whey protein concentrate (Experimental): 2 servings daily
  Serving information:
  * 192 kcal
  * 4.6 g fat
  * 12.2 g carbohydrate
  * 25.4 g protein (2.9 g L-leucine)
  Interventions: Dietary Supplement: Hydrolyzed whey protein concentrate
- Soy protein concentrate (Experimental): 2 servings daily
  Serving information:
  * 266 kcal
  * 4.5 g fat
  * 17.2 g carbohydrate
  * 39.2 g protein (2.9 g L-leucine)
  Interventions: Dietary Supplement: Soy protein concentrate

INTERVENTIONS:
Dietary Supplement: Placebo — Supplementation twice daily (1 serving dose per consumption) of maltodextin while engaging in resistance training 3 times per week for a 12-week period. Supplementation occurred during training and non-training days.
  Arms: Placebo
Dietary Supplement: L-leucine + maltodextrin — Supplementation twice daily (1 serving dose per consumption) of L-leucine + maltodextin while engaging in resistance training 3 times per week for a 12-week period. Supplementation occurred during training and non-training days.
  Arms: L-leucine + maltodextrin
Dietary Supplement: Whey protein concentrate — Supplementation twice daily (1 serving dose per consumption) of whey protein concentrate while engaging in resistance training 3 times per week for a 12-week period. Supplementation occurred during training and non-training days.
  Arms: Whey protein concentrate
Dietary Supplement: Hydrolyzed whey protein concentrate — Supplementation twice daily (1 serving dose per consumption) of hydrolyzed whey protein concentrate while engaging in resistance training 3 times per week for a 12-week period. Supplementation occurred during training and non-training days.
  Arms: Hydrolyzed whey protein concentrate
Dietary Supplement: Soy protein concentrate — Supplementation twice daily (1 serving dose per consumption) of soy protein concentrate while engaging in resistance training 3 times per week for a 12-week period. Supplementation occurred during training and non-training days.
  Arms: Soy protein concentrate

SUMMARY:
The purpose of this study was to determine the effects of L-leucine (LEU) or different protein supplements standardized to LEU (~3.0 g/serving) on changes in body composition, strength, and histological attributes in skeletal muscle and adipose tissue. Seventy-five untrained, college-aged males (mean±SE; age=21±1 yr, body mass=79.2±0.3 kg) were randomly assigned to an isocaloric, lipid-, and organoleptically-matched maltodextrin placebo (PLA, n=15), LEU (n=14), whey protein concentrate (WPC, n=17), whey protein hydrolysate (WPH, n=14), or soy protein concentrate (SPC, n=15) group. Participants performed whole-body resistance training three days per week for 12 weeks while consuming supplements twice daily. Skeletal muscle and subcutaneous (SQ) fat biopsies were obtained at baseline (T1) and ~72 h following the last day of training (T39). Tissue samples were analyzed for changes in type I and II fiber cross sectional area (CSA), non-fiber specific satellite cell count, and SQ adipocyte CSA. On average, all supplement groups including PLA exhibited similar training volumes and experienced statistically similar increases in total body skeletal muscle mass determined by dual x-ray absorptiometry (+2.2 kg; time p=0.024) and type I and II fiber CSA increases (+394 µm2 and +927 µm2; time p<0.001 and 0.024, respectively). Notably, all groups reported increasing Calorie intakes ~600-800 kcal/d from T1 to T39 (time p<0.001), and all groups consumed at least 1.1 g/kg/d of protein at T1 and 1.3 g/kg/d at T39. There was a training, but no supplementation, effect regarding the reduction in SQ adipocyte CSA (-210 µm2; time p=0.001). Interestingly, satellite cell counts within the WPC (p<0.05) and WPH (p<0.05) groups were greater at T39 relative to T1. In summary, LEU or protein supplementation (standardized to LEU content) does not provide added benefit in increasing whole-body skeletal muscle mass or strength above PLA following 3 months of training in previously untrained college-aged males that increase Calorie intakes with resistance training and consume above the recommended daily intake of protein throughout training. However, whey protein supplementation increases skeletal muscle satellite cell number in this population, and this phenomena may promote more favorable training adaptations over more prolonged periods.

DETAILED DESCRIPTION:
OVERALL STUDY DESIGN The study design implemented was double-blinded and placebo-controlled. Likewise, guidelines established by the CONSORT Transparent Reporting of Trials established in 2010 (www.consort-statement.org) were followed. Participants were encouraged to refrain from rigorous physical activity for 4-5 days prior to baseline testing (T1). For T1, participants were instructed to report to the laboratory in a well-hydrated, 4-hour fasted state whereby they were subjected to the following assessments: a) urine specific gravity, b) height and body mass, c) body composition using dual-energy X-ray absorptiometry (DXA) (General Electric Lunar Prodigy enCORE, software version 10.50.086; Madison, WI, USA), d) vastus lateralis thickness using ultrasonography (General Electric LOGIQ S7 Expert; Chicago, IL, USA), e) venipuncture, f) percutaneous skeletal muscle biopsy collection from the vastus lateralis, and g) a percutaneous SQ fat biopsy from the gluteal region. Two to three days following T1, subjects reported back to the laboratory in a 4-hour fasted state for a second visit (T2) whereby maximal force production capacity was assessed using an isometric mid-thigh pull (IMTP) test, lower body strength was assessed using a three repetition maximum (3-RM) squat, and upper body strength was assessed using a 3-RM bench press. Additionally, during T2, subjects were familiarized with all lifts that were to be performed during the training intervention. Following T2, subjects engaged in 12 weeks of resistance training and supplementation. The last training bout (T38) consisted of IMTP as well as squat and bench press 3-RM re-assessments in a 4-hour fasted state. Seventy two hours following T38, subjects reported back to the laboratory in a 4-hour fasted state for post-testing (T39) which consisted of all body composition, and blood and biopsy collection procedures noted for T1.

RESISTANCE TRAINING PROTOCOL For visits 3-37 (T3-T37), a daily undulating periodization training model was employed over the 12-week training period given that this model has been shown to be more beneficial in eliciting greater increases in strength and hypertrophy than traditional linear training models. Specifically, participants were instructed to perform free-weighted barbell squats, bench press, deadlifts, and bent-over-rows for 4 sets of 10 repetitions (Monday or Tuesday), 6 sets of 4 repetitions (Wednesday or Thursday), and 5 sets of 6 repetitions (Friday or Sunday). Immediately following each completed set, a rating of perceived exertion score was acquired from each participant (scale: 1-10) in order to monitor and progress each participant accordingly while minimizing the potential risk of injury. The RPE scale was described to participants as the remaining number of repetitions that the participant would be able to complete while employing good technique (i.e., 1 = 9 remaining repetitions in reserve, 10 = 0 remaining repetitions in reserve). More information on relative training intensities and progression can be found in Table 1. Participants were instructed to attend all 36 resistance training sessions throughout the duration of the study, but those that missed more than 4 sessions were not included in the analysis due to lack of training compliance. All participants were supervised by laboratory personnel for each training session to ensure that proper lifting technique was executed, and training volumes for each session were recorded.

SUPPLEMENTATION PROTOCOL As stated above, participants were assigned to ingest either a PLA, LEU, WPC, WPH, or SPC supplement throughout the training intervention. On training days (T3-T37), participants consumed an individually-packaged serving in ~500 ml of tap water immediately following each training session under direct observation of the study personnel. Additionally, participants were instructed to consume an individual serving within 30 min prior to bedtime. On non-training days, participants were instructed to consume an individual serving between a meal of their choosing and 30 min prior to bedtime. Supplements were separated into individual ready-made supplement-coded packets for daily consumption, and participants were given a 3-week supply. Study personnel collected and counted empty packets from each participant every 3 weeks before the next 3-week supply was distributed. Participants that did not consume >80% were not included in the analysis due to lack of compliance. Each supplement, except PLA, was formulated to provide ~3 g of leucine, per serving. Furthermore, each supplement was formulated to yield similar amounts of total energy (kcal) and fat (g), and was double-blinded to laboratory personnel and participants for group, appearance, taste, texture, and packaging. The WPC supplement was formulated using an agglomerated, 80% WPC (Hilmar™ 8010, Hilmar Ingredients; Hilmar, CA, USA). The WPH supplement was formulated using an agglomerated, partially hydrolyzed [12.5% degree of hydrolysate (12.5% DH), yielding approximately 67% of peptides as <5 kilodaltons (kDa) in molecular weight] 80% whey protein concentrate (Hilmar™ 8360, Hilmar Ingredients); SPC used an agglomerated, 80% soy protein concentrate (ALPHA® 5812, Solae, LLC; St. Louis, MO, USA); LEU used an agglomerated, L-Leucine (L-Leucine USP, Glambia Nutritionals; Carlsbad, CA, USA) and non-GMO, corn-derived maltodextrin (MALTRIN®-M100; Grain Processing Corporation; Muscantine, IA, USA); and, the PLA group was formulated using maltodextrin (MALTRIN®-M100; Grain Processing Corporation). All five supplements were manufactured at JW Nutritional, LLC (Allen, TX, USA), a United States Food and Drug Administration cGMP-compliant facility independently audited and pre-qualified by Obvium*Q, LLC (Phoenix, AZ, USA), a GMP regulatory compliance firm. Personnel at JW Nutritional, LLC and a third-party organization (Lockwood, LLC; Draper, UT, USA) formulated and maintained blinding of groups, and each supplement was assigned a randomly generated item number. Manufacturing batch records for production of each of the five supplements were reviewed by a trained, independent expert in dietary supplement quality control and assurance before approval for use within the present study. All supplements were independently validated for nutritional facts and total amino acids using validated, approved methods at Covance Laboratories, Inc. (Madison, WI, USA), a pre-qualified third-party analytical laboratory, and results reviewed by a third-party organization (Lockwood, LLC) prior to the supplements being approved for use within the present study. Once analysis was complete, a third-party organization (Lockwood, LLC) representative not involved in the study released the code for all treatments.

ELIGIBILITY:
Inclusion Criteria:

1. are between the ages of 19-35 and have a body mass index (body mass in kilograms/ height in meters^2) between 23-30
2. are apparently healthy and do not have any known illnesses that are contraindicated for exercise (i.e., hypertension, arrhythmias, or cardiopulmonary diseases), or are not taking medications for these diseases
3. have not engaged in lower-body weight training over the past 12 months; this means less than one training session per every two weeks
4. have not engaged in lower-body endurance training over the past 12 months; this means that the participant has not run more than 10 miles per week or road-biked/swam more than 2 days per week
5. have not consumed nutritional supplements two months prior to the study including hormone boosters, protein supplements, amino acid supplements and/or creatine monohydrate
6. are not regular tobacco users, or haven't been over the past 12 months
7. do not have any blood clotting issues and/or are on blood-thinning agents or medications

Exclusion Criteria:

1. are not between the ages of 19-35 or have a body mass index (body mass in kilograms/ height in meters^2) outside the range of 23-30
2. have any known illnesses that are contraindicated for exercise (i.e., hypertension, arrhythmias, or cardiopulmonary diseases), or are not taking medications for these diseases
3. have engaged in lower-body weight training over the past 12 months
4. have engaged in lower-body endurance training over the past 12 months
5. have consumed nutritional supplements two months prior to the study including hormone boosters, protein supplements, amino acid supplements and/or creatine monohydrate
6. are tobacco users
7. have any blood clotting issues and/or are on blood-thinning agents or medications

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 89 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Index of skeletal muscle hypertrophy | Pre- and post-intervention assessments (12-week seperation between assessments)
  Whole-body dual x-ray absorptiometry scan for lean body mass assessment (units in kilograms)

SECONDARY OUTCOMES:
Index of muscle hypertrophy at the cellular level | Pre- and post-intervention assessments (12-week seperation between assessments)
  Muscle fiber cross-sectional area assessment from biopsy specimens via histological methods (units in micrometers-squared)
Index of whole-body adiposity | Pre- and post-intervention assessments (12-week seperation between assessments)
  Whole-body dual x-ray absorptiometry scan for fat mass assessment (units in kilograms)
Index of cellular adiposity | Pre- and post-intervention assessments (12-week seperation between assessments)
  Subcutaneous fat cell cross-sectional area assessment of biopsy specimens via histological methods (units in micrometers-squared)

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing can be achieved by contacting the PI at mdr0024@auburn.edu.